CLINICAL TRIAL: NCT00084916
Title: A Phase II Study Of CCI-779 In Patients With Relapsed Or Refractory Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, Or Chronic Myeloid Leukemia In Blastic-Phase
Brief Title: CCI-779 in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Myelodysplastic Syndromes, or Chronic Myelogenous Leukemia in Blastic Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02589; MDA-2003-0830; N01CM62202 (NIH); CDR0000367093 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy such as CCI-779 work in different ways to stop cancer cells from dividing so they stop growing or die. This phase II trial is studying how well CCI-779 works in treating patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, or chronic myelogenous leukemia in blastic phase

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the activity of CCI-779 in patients with relapsed or refractory acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndromes, or chronic myelogenous leukemia in blastic phase.

II. Correlate the effect of this drug with altered mitochondrial respiration in the leukemia cells of these patients.

OUTLINE: Patients are stratified according to disease (acute myeloid leukemia, myelodysplastic syndromes, chronic myelogenous leukemia in blastic phase [CML-BP] non-lymphoid vs acute lymphoblastic leukemia, CML-BP lymphoid).

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 24-74 patients (12-37 per stratum) will be accrued for this study within 8-46 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Myelodysplastic syndromes

    * Refractory anemia with excess blasts [RAEB]
    * RAEB in transformation
    * Chronic myelomonocytic leukemia in transformation with ≥ 10% peripheral blood/bone marrow blasts
  * Chronic myelogenous leukemia in blastic phase
* Disease status must meet 1 of the following criteria:

  * Primary resistant disease (i.e., failed to achieve a complete response [CR] to a prior standard induction regimen)
  * Relapsed disease after achieving a CR
* Documented failure to most recent cytotoxic regimen
* No other potentially curative options
* No known CNS disease
* Performance status - ECOG 0-2
* SGOT or SGPT < 3 times upper limit of normal*
* Bilirubin ≤ 2 mg/dL*
* Creatinine ≤ 2 mg/dL (unless due to organ leukemic involvement)
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to CCI-779
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No AIDS-defining disease

  * HIV positive allowed if CD4 counts normal
* No other concurrent uncontrolled illness
* No concurrent prophylactic hematopoietic colony-stimulating factors
* More than 2 weeks since prior cytotoxic chemotherapy (except hydroxyurea) and recovered
* More than 2 weeks since prior radiotherapy and recovered
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-04; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Response rate of 20% | Up to 3 years
  The 95% confidence intervals should be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giles, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States